CLINICAL TRIAL: NCT00745628
Title: Cross-Sectional Investigation of Secondary Prevention on Coronary Heart Disease and Generalization of Standardized Secondary Prevention in Chinese Coronary Heart Disease Patients
Brief Title: Chinese Cohort Study of Coronary Heart Disease
Acronym: CCS-CHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: YHuo,director, Peking University First Hospital
Other Study IDs: 2006BAI01A02-08
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Heart Diseases
Keywords: coronary heart disease; secondary prevention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Construction of coronary heart disease cohort of more than 10000 patients in China. Investigation on current situation of secondary prevention of CHD will be carried out and the effect of physician training and patient education will be evaluated.

DETAILED DESCRIPTION:
More than 40 hospitals of 16 provinces will enroll patients for this study. The study will include patients with diagnosed coronary heart disease. Investigators and all the physicians who will involve in daily care of CHD patients will have a brief training on guideline of secondary prevention in CHD and take a test on that. Questionnaires are used to evaluate patient's cognition of their diseases and knowledge on coronary heart disease. Patient education will be carried out during a 2 years follow up of all the patient enrolled before they are required to fill out another questionnaire. Physicians will also take a second test on secondary prevention of CHD at that time. Patients will take blood lipids and glucose test according to their physician's requirement.The effect of physician training and patient education will be evaluated by comparing the results of questionnaires and tests at the beginning of the study and in the end of the 2 years follow up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed coronary heart disease
* Confirmed by coronary angiography;
* Diagnosed myocardial infarction;
* Typical symptom of ischemic chest pain with positive stress test;
* Willing to sign an inform consent.

Exclusion Criteria

* Patients won't sign an inform consent or will not comply with the follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Hong, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China